CLINICAL TRIAL: NCT03889977
Title: The Effect of Resistance Exercise on Postprandial Hyperglycemia in Patients With B-thalassemia Exhibiting Resistance to Insulin (Type II Diabetes and Prediabetes)
Brief Title: Resistance Exercise on Postprandial Hyperglycemia in Patients With B-thalassemia Exhibiting Resistance to Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-Thalassemia ResEx Glucose
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Beta-Thalassemia; Insulin Resistance; PreDiabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — beta-Thalassemia; Insulin Resistance; Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Resistance exercise 45 min following breakfast
  Interventions: Other: Resistance exercise
- Control (No Intervention): No exercise (resting) following breakfast

INTERVENTIONS:
Other: Resistance exercise — 2 major muscle groups (lower extremity, chest)
  Arms: Exercise

SUMMARY:
It is known that postprandial hyperglycemia increases the cardiometabolic risk in both diabetic and non-diabetic patients. Moreover, there is insufficient data on the effectiveness of exercise on preventing Type II diabetes mellitus in individuals with insulin resistance and prediabetes. This study aims to examine the effectiveness of resistance exercise in limiting postprandial hyperglycemia and the necessity of prescribing medication particularly in patients with beta-thalassemia and insulin resistance.

DETAILED DESCRIPTION:
Type II diabetes mellitus is a condition characterized by chronic hyperglycemia due to insufficient insulin production and action and tissue resistance to insulin. Pre-diabetes is also characterized by elevated levels of blood glucose, but not so high as those in diabetes.

Existing studies have shown that postprandial hyperglycemia is associated with an increased risk for complications of diabetes, both microvascular and macrovascular, as it contributes to the deficiency of β-pancreatic cells and endothelial dysfunction to a much greater extent than glycosylated hemoglobin (HbA1c) and fasting glucose.

The main problem in glycemic control is the glucose peak 1-2 hours after the meal. Therefore, there is a need to investigate whether postprandial exercise can help solve this problem.

Βeta-thalassemia is a group of heterogeneous hereditary anemias characterized by decreased or no production of beta-chain hemoglobin, resulting in inefficient erythropoiesis. The three main phenotypes are: a) major b) intermediate and c) heterozygous beta-thalassemia. Major thalassemia occurs in the first 2 years of life with severe anemia and requires systemic transfusions. The intermediate appears later and usually does not need transfusions. The heterozygote is asymptomatic, but some carriers may experience mild anemia. Beta-thalassemia is inherited in an autosomal recessive manner. Patient survival has increased significantly in recent years due to systemic transfusions and early treatment of disease complications. However, multiple transfusions result in the accumulation of large quantities of iron, which is toxic to pancreatic beta cells. Both decreased insulin production and decreased tissue sensitivity to insulin occur and result in pre-diabetes or Type II diabetes.

Regarding the effect of exercise on diabetic patients, it is confirmed that it reduces both the blood glucose concentration and hyperglycemia during the day. Resistance exercise increases heat production and oxygen consumption by the muscles, thus increasing metabolic activity and glucose uptake by these muscles. In addition, resistance exercise improves glycemic control without causing hypoglycemia and without affecting fasting glucose. Thus, the aim of this study is examine the effectiveness of resistance exercise in limiting postprandial hyperglycemia in patients with beta-thalassemia and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Beta-Thalassemia
* Diagnosed with prediabetes or type II diabetes

Exclusion Criteria:

* Heart failure
* Hypertension
* Muscular, neuromuscular, bone disorders
* Muscular, bone or other injuries that do not allowed safe participation to exercise

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose | Pre-breakfast (fasting glucose), 45 min post-breakfast (before exercise), immediately post-exercise, 1 hour post-exercise, 2 hours post-exercise, 24 hours post-exercise
  Concentration of blood glucose will be measured in serum
Changes in blood insulin | Pre-breakfast (fasting glucose), 45 min post-breakfast (before exercise), immediately post-exercise, 1 hour post-exercise, 2 hours post-exercise, 24 hours post-exercise
  Concentration of blood insulin will be measured in serum
Changes in blood triglycerides | Pre-breakfast (fasting glucose), 45 min post-breakfast (before exercise), immediately post-exercise, 1 hour post-exercise, 2 hours post-exercise, 24 hours post-exercise
  Concentration of blood triglycerides will be measured in serum

SECONDARY OUTCOMES:
Body mass | At the baseline and before each trial
  Body mass (kg) will be measured with Beam Balance-Stadiometer (SECA, Vogel & Halke, Hamburg, Germany)
Body height | At the baseline
  Body height (m) will be measured with Beam Balance-Stadiometer (SECA, Vogel & Halke, Hamburg, Germany)
Body fat | Before each trial
  Body fat (kg and percentage) will be measured with Dual-emission X-ray absorptiometry (GE Healthcare, Lunar DPX-NT)
Resting heart rate | At the baseline and before each trial
  Resting heart rate (beats per minute) will be monitored using Team Polar (Polar Electro Oy, Kempele, Finland)
Heart rate during exercise | During exercise in each trial
  Heart rate (beats per minute) will be monitored using continuous heart rate measurements (Team Polar, Polar Electro Oy, Kempele, Finland)
Changes in total antioxidant capacity | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of total antioxidant capacity will be measured in serum
Changes in reduced glutathione (GSH) | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of GSH will be measured in erythrocyte lysate
Changes in catalase | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of catalase will be measured in erythrocyte lysate
Changes in uric acid | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of uric acid will be measured in serum
Changes in protein carbonyls | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of protein carbonyls will be measured in plasma
Changes in substances that react with thiobarbituric acid (TBARS) | Pre-breakfast (fasting glucose), immediately post-exercise, 24 hours post-exercise
  Concentration of TBARS will be measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Stamperna, MD, Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece